CLINICAL TRIAL: NCT06444542
Title: Understanding Patient Preference on Colorectal Cancer Screening Options
Brief Title: Understanding Patient Preference on Colorectal Cancer Screening Options-PSU
Acronym: U-Screen
Status: Recruiting | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Guardant Health, Inc. (Industry); HealthLinc, Inc (Unknown); PCC Community Wellness Center (Unknown)
Responsible Party: Principal Investigator, Karen Kim, Dean at Penn State College of Medicine, Milton S. Hershey Medical Center
Other Study IDs: STUDY00023853
Record Dates: First submitted 2024-05-14; First posted 2024-06-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Guardant Shield — Blood-based colorectal cancer screening

SUMMARY:
There are significant barriers to colorectal cancer screening within underserved populations due to the cost, accessibility, and acceptability of screening methods. Patient-friendly approaches that minimize stress and discomfort for the patient are needed to enhance screening compliance and achieve an early diagnosis. The primary aim of this study is to examine whether the availability of a blood-based screening option, which can be done at the point of service and is familiar to patients, will improve patient compliance to recommended CRC screening

DETAILED DESCRIPTION:
Scientific Background and Gaps Colorectal cancer (CRC) is the third most common cancer type and the second leading cause of cancer death in the United States. The lethal nature of CRC is attributable to its being largely asymptomatic during the early stages and the lack of curative treatment options for patients with progressive disease. Early detection by screening significantly reduces mortality from CRC; however, many people are not up to date with screening, with overall screening rates under 70%. Furthermore, about a quarter of age-eligible adults (27.1 million) have never been screened for CRC. A recent study found that not being up to date with screening was associated with an approximate 3-fold risk for CRC-related mortality. Despite many years of effort and funding support, CRC screening rates have plateaued, with a considerable segment of the population remaining unscreened. The percentage of age-eligible adults who were up to date with CRC screening only increased by 1.4% (4.2 million) from 67.4% in 2016 to 68.8% in 2018. Compliance with CRC screening is particularly poor among medically underserved populations, including those with low income and racial/ethnic minority populations. There are significant barriers to screening within underserved populations due to the cost, accessibility, and acceptability of screening methods. To date, there are many well-established CRC screening modalities and can include invasive and non-invasive options that detect both polyps and cancer or cancer alone. Colonoscopy is considered the gold standard for CRC screening and remains the dominant screening modality in the U.S. However, due to the invasiveness, perception of discomfort and embarrassment, logistical challenges (e.g., lack of transportation, time off of work), cost, and potential risks, the uptake of colonoscopy is low. For patients unwilling to screen with colonoscopy, non-invasive stool-based testing can shift CRC detection to earlier and more curable stages. However, the compliance of stool-based testing is suboptimal due to the cultural stigma surrounding sample collection techniques and the inconvenience of returning the kit for testing. Increasing patient compliance and adherence to screening is critical to improving CRC outcomes. Patient-friendly approaches that minimize stress and discomfort for the patient are needed to enhance screening compliance and achieve an early diagnosis. A blood-based screening option can improve CRC screening uptake and adherence at FQHCs, and, ultimately, eliminate unnecessary cancer disparities.

Previous Data Patient compliance is a major barrier to achieving universal screening. Blood-based testing can offer an alternative for patients who fail to comply with other screening modalities. Blood tests are non-invasive compared to colonoscopy, and individuals are more willing to have a blood test than take a stool sample at home. In a cross-sectional survey of 100 individuals, 91% ranked a blood-based test as their first or second choice of screening (58% for the first choice, 10% tied, and 23% for the second choice) compared with colonoscopy, sigmoidoscopy, or stool-based tests. Furthermore, over two-thirds of minority respondents (n=62) chose a blood-based screening test as their first choice for future screening. Blood-based screening test also presents an opportunity to overcome challenging barriers, such as transportation and time off from work, limiting screening participation.

Study Rationale A key to improving screening participation is patient acceptance of the testing method. Indeed, all the screening modalities have benefits over time, and compliance to testing is essential for successful screening. A blood-based screening test can easily be part of a routine clinic visit and the patient can complete the test while is still at the clinic. Patients are accustomed to providing blood samples for other screening tests, such as cholesterol screening and the use of blood-based CRC screening test is likely more in line with a patient's expectations of medical care. On January 19, 2021, the Centers for Medicare and Medicaid Services announced that the blood-based biomarker test is an appropriate CRC screening once every 3 years for Medicare patients when performed in a CLIA-certified laboratory, ordered by a treating physician, and the blood-based biomarker screening test has a sensitivity greater than or equal to 74% and a specificity greater than or equal to 90% in the detection of CRC.

The last decades have seen many discovery studies identifying promising biomarkers of CRC. Improving testing methods for blood-based CRC testing have been developed and implemented in clinical settings as well. The first blood-based CRC screening test, SEPT9 DNA (Epi proColon), was approved by the FDA in 2016 for persons at average risk for CRC who have chosen not to undergo screening by existing guideline-recommended methods. This study will offer a lab-developed Guardant SHIELD blood-based CRC screening test to patients who failed to complete a stool-based screening test or a colonoscopy six months after receiving an order from their providers. The Guardant SHIELD blood-based screening test will be free to the patients with an order from their providers. The Guardant SHIELD test is a multimodal blood-based colorectal neoplasia detection assay incorporating ctDNA (circulating tumor DNA) assessment of somatic mutations and tumor-derived methylation and fragmentomic patterns to maximize early-stage CRC detection sensitivity. Overall, the Guardant SHIELD blood-based test has a CRC sensitivity of 91% and a specificity of 94%, meeting the Centers for Medicare and Medicaid Services requirement (74% for sensitivity and 90% for specificity). All the blood samples collected in this study will be processed at the CLIA-certified Guardant Health Laboratory.

Compliance by age-eligible patients is essential to the success of any screening program. However, the acceptance by health care providers and the health care system is also critical, and especially colonoscopy remains the dominant modality for CRC in the U.S. Applying the current state of research evidence to health care involves fostering the adoption, implementation, spread, and sustainability of new evidence-based interventions to care. Furthermore, transferring effective interventions into real-world settings and maintaining them is a complicated, long-term process that requires complex phases of intervention diffusion. In this study, we will examine the inclusion of a blood-based screening option to increase patient compliance with CRC screening while developing implementation strategies to facilitate the adoption of a new blood-based screening test at primary care clinics.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, participants must meet all the following criteria:

1. Between 45-75 years of age
2. Language Proficiency: participants must be fluent in English or Spanish
3. Have an average risk for colorectal cancer
4. Be a patient at one of our partner FQHCs
5. Received a screening order (either using a stool-based test or colonoscopy) six months ago and failed or refused to complete the screening test
6. Able and willing to provide a blood sample per protocol

Exclusion Criteria:

Participants will be excluded from enrolling in the study if they meet any of the following:

1. Family history

   * One first-degree relative diagnosed with CRC or advanced adenoma at age <60 years
   * Two first-degree relatives diagnosed with CRC or advanced adenoma at any age
   * Known hereditary gastrointestinal cancer syndromes, such as Lynch Syndrome or Familial Adenomatous and Polyposis (FAP)
2. Personal History

   * Participants who do not speak either Spanish or English
   * History of CRC or adenoma
   * History of cancers
   * History of inflammatory bowel disease, including chronic ulcerative colitis and Crohn's disease
   * Have a recorded up to date CRC screening
   * Blood product transfusion in the past 120 days
   * A medical condition which, in the opinion of the patient's health provider, should preclude enrollment in the study

Ages: 45 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who failed to complete a stool-based screening test or a colonoscopy six months after receiving an order from their providers
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient preference for a blood-based screening option | 2023-2025
  We will ask participants the following survey question: "Will you prefer to use the blood-based screening test for future colorectal cancer screening?" Response options range from 0 to 10 where 0 is "not at all" and 10 is "very much". We will split the response options at the median and categorize the measure into a "yes/no" response.

SECONDARY OUTCOMES:
Adoption rate | 2023-2025
  This study will monitor the adoption rates for Guardant SHIELD blood-based screening over time and how long it takes to achieve 2.5%, 16%, and 50% adoption rates (adoption rate = the number of new users / total number of potential users). We will monitor the adoption rate quarterly. In addition, we will also monitor the intensity of use.
  This study will monitor the adoption rates for Guardant SHIELD blood-based screening over time and how long it takes to achieve 2.5%, 16%, and 50% adoption rates (adoption rate = the number of new users / total number of potential users). We will monitor the adoption rate quarterly. In addition, we will also monitor the intensity of use

CONTACTS AND LOCATIONS:
Overall Officials: Karen E. Kim, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No